CLINICAL TRIAL: NCT01301092
Title: A Study to Evaluate the Safety, Tolerability, and Absolute Bioavailability of Subcutaneous LY2189265
Brief Title: A Study to Compare the Concentrations of LY2189265 After Different Methods of Administration to Healthy Volunteers.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 13989; H9X-MC-GBDR (Other: Eli Lilly and Company)
Record Dates: First submitted 2011-02-18; First posted 2011-02-23 (Estimated); Results first posted 2014-10-07 (Estimated); Last update posted 2014-10-07 (Estimated); Status verified 2014-10

CONDITIONS: Diabetes Mellitus, Type II
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dulaglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Part A: LY2189265 intravenous (Experimental): Single intravenous (IV) dose, starting at 0.1 milligrams (mg) of LY2189265. Dose may be increased to 0.2 mg or decreased to 0.05 mg for subsequent patients, dependent on safety assessments of the first 3 patients.
  Interventions: Biological: LY2189265
- Part B: LY2189265 subcutaneous, intravenous (Experimental): Patients are randomized to 2 sequences of 2 treatments. Single 1.5 mg subcutaneous (SC) dose of LY2189265 in Period 1; single intravenous (IV) dose of LY2189265 (determined by Part A IV arm data) in Period 2 or vice versa. There is a washout period of at least 4 weeks between dosing periods.
  Interventions: Biological: LY2189265
- Part C: LY2189265 subcutaneous, intramuscular (Experimental): Patients are randomized to 2 sequences of 2 treatments. Single 0.75 mg subcutaneous (SC) dose of LY2189265 in Period 1; single 0.75 mg intramuscular (IM) of LY2189265 in Period 2 or vice versa. There is a washout period of at least 4 weeks between dosing periods.
  Interventions: Biological: LY2189265

INTERVENTIONS:
Biological: LY2189265 — administered intravenous, subcutaneous or intramuscular

SUMMARY:
LY2189265 is an investigational drug being developed for the treatment of type 2 diabetes mellitus. This study will compare the concentrations of LY2189265 using different methods of administration: subcutaneous (or SC- an injection just under the skin), intravenous (or IV - into a vein in the arm) and intramuscular (IM - into the muscle of the left thigh). The purpose of this study is to look at how much of the drug gets into the blood stream and how long it takes the body to get rid of it when given by the methods above. The study is divided into three parts, Part A, B and C. Volunteers will only be able to participate in one part. All Participants in Part A will receive a single IV dose of up to 0.1 milligram (mg). Participants in Part B will be given drug twice by IV and an SC injection (1.5 mg). Part B of the study will occur after Part A because the dose of IV drug will depend on the results of Part A. Part B of the study may not occur if the volunteers in Part A do not tolerate the drug. Participants in Part C will also be given drug twice by an SC injection and an IM injection, both doses will be 0.75 mg.

ELIGIBILITY:
Inclusion Criteria:

* Are overtly healthy males or females, as determined by medical history and physical examination.
* Male subjects with female partners of child-bearing potential, or partners who are pregnant or breastfeeding, agree to use a reliable method of contraception from the time of the first dose until 3 months after the last dose of investigational product, as determined by the investigator. The method may be one of the following: condom with spermicidal agent, male subject sterilization, true abstinence (which is in line with the subject's usual lifestyle choice; withdrawal or calendar methods are not considered acceptable).
* Female subjects not of child-bearing potential (that is, are postmenopausal or permanently sterilized [for example, tubal occlusion, hysterectomy, bilateral salpingectomy]). Such subjects will not be required to use contraception but must test negative for pregnancy at the time of enrollment. Postmenopausal is defined as at least 1 year post cessation of menses (without an alternative medical cause) with follicle stimulating hormone (FSH) greater than or equal to 40 milli-international units per milliliter (mIU/mL).
* Female subjects who have undergone sterilization by tubal ligation: agree to use a condom in conjunction with spermicidal gel, foam, cream, film or suppository from the time of screening until 3 months after the last dose of investigational product. Such subjects must also test negative for pregnancy at the time of enrollment.
* Have a body mass index (BMI) of between 23.0 and 35.0 kilogram/square meter (kg/m²), inclusive.
* Have clinical laboratory test results within normal reference range for the population or investigator site, or results with acceptable deviations that are judged to be not clinically significant by the investigator.
* Have normal sitting blood pressure and pulse rate as determined by the investigator, or with changes compatible with their age.
* Have venous access sufficient to allow for blood sampling and/or IV administration of investigational product as per the protocol.
* Are reliable and willing to make themselves available for the duration of the study and are willing to follow study procedures.
* Have given written informed consent approved by Lilly and the ethical review board (ERB) governing the site.

Exclusion Criteria:

* Are currently enrolled in, or discontinued within the last 30 days from, a clinical trial involving an investigational drug or device, or are concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study.
* Are women of child bearing potential
* Have known allergies to Glucagon-like peptide-1 (GLP-1)-related compounds including LY2189265.
* Are persons who have previously completed or withdrawn from this study or any other study investigating LY2189265.
* Have an abnormality in the 12-lead Electrocardiogram (ECG) that, in the opinion of the investigator, increases the risks associated with participating in the study.
* Have a history or presence of gastrointestinal disorder (including pancreatitis [history of chronic pancreatitis or idiopathic acute pancreatitis] or gall bladder disease), or gastrointestinal disease that impacts gastric emptying (GE) (for example, gastric bypass surgery, pyloric stenosis) or could be aggravated by GLP analogs (for example, esophageal reflux). Subjects having had cholecystolithiasis (removal of gall stones), cholecystectomy (removal of gall bladder) and/or appendectomy in the past with no further sequelae may be included in the study at the discretion of the screening physician.
* Have a history or presence of significant active neuropsychiatric disease
* Regularly use known drugs of abuse and/or show positive findings on urinary drug screening.
* Show evidence of human immunodeficiency virus (HIV) and/or positive human HIV antibodies.
* Show evidence of hepatitis C and/or positive hepatitis C antibody.
* Show evidence of hepatitis B and/or positive hepatitis B surface antigen.
* Are women with a positive pregnancy test or women who are lactating.
* Use or intend to use over-the-counter medication other than paracetamol within 7 days prior to dosing or prescription medication (with the exception of vitamin/mineral supplements and/or hormone replacement therapy and/or thyroid replacement therapy) within 14 days prior to dosing.
* Have donated blood of more than 500 mL within the last month.
* Are subjects who have an average weekly alcohol intake that exceeds 21 units per week (males) and 14 units per week (females), (1 unit = 12 ounce [oz] or 360 mL of beer; 5 oz or 150 mL of wine; 1.5 oz or 45 mL of distilled spirits), or are unwilling to stop alcohol consumption from at least 24 hours prior to screening and each dose, and while resident at the clinical research unit (CRU).
* Are subjects who smoke more than 10 cigarettes per day, are unwilling to refrain from smoking on the day of LY2189265 administration and while resident.
* Are subjects who, in the opinion of the investigator, are in any way unsuitable to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-02; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Evansville, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Part A: LY2189265 Intravenous: Single 0.1-milligram (mg) intravenous (IV) dose of LY2189265.
- Part B: LY2189265 Subcutaneous, Intravenous: Participants were randomized to 2 sequences of 2 treatments. Single 1.5-mg subcutaneous (SC) dose of LY2189265 in Period 1; single 0.1-mg intravenous (IV) dose of LY2189265 in Period 2 or vice versa. There was a washout period of at least 4 weeks between dosing periods.
- Part C: LY2189265 Subcutaneous, Intramuscular: Participants were randomized to 2 sequences of 2 treatments. Single 0.75-mg subcutaneous (SC) dose of LY2189265 in Period 1; single 0.75-mg intramuscular (IM) of LY2189265 in Period 2 or vice versa. There was a washout period of at least 4 weeks between dosing periods.
Period: Overall Study
Arm/Group | Part A: LY2189265 Intravenous | Part B: LY2189265 Subcutaneous, Intravenous | Part C: LY2189265 Subcutaneous, Intramuscular
Started | 6 | 16 | 8
Completed | 6 | 16 | 7
Not Completed | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Part A: LY2189265 Intravenous: Single 0.1 milligram (mg) intravenous (IV) dose of LY2189265
- Total: Total of all reporting groups
Arm/Group | Part A: LY2189265 Intravenous | Part B: LY2189265 Subcutaneous, Intravenous | Part C: LY2189265 Subcutaneous, Intramuscular | Total
Number analyzed (Participants) | 6 | 16 | 8 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.0 (13.1) | 42.3 (15.0) | 45.6 (16.6) | 44.10 (14.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 3 | 10
  Male | 3 | 12 | 5 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 5 | 16 | 8 | 29
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 3 | 5
  White | 6 | 14 | 5 | 25
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 16 | 8 | 30

OUTCOME MEASURES:

1. Primary Outcome: Dose Normalized Area Under the Concentration Time Curve (AUC) of LY2189265: Subcutaneous (SC) to Intravenous (IV)
Description: AUC is AUC from time zero to infinity. The results presented are Geometric Least Squares (LS) Mean. LS Mean values were controlled for participants, sequence, treatment, period and random error.
Time Frame: Predose up to 336 hours postdose
Population: Participants in Part B who had pharmacokinetic (PK) data.
Measure: Geometric Mean (90% Confidence Interval); unit: nanograms*hour/milliliter/milligram
Groups:
- Part B: LY2189265 Subcutaneous: Single 1.5 mg-subcutaneous (SC) dose of LY2189265 in Period 1 or 2
- Part B: LY2189265 Intravenous: Single 0.1-mg intravenous (IV) dose of LY2189265 in Period 1 or 2
Arm/Group | Part B: LY2189265 Subcutaneous | Part B: LY2189265 Intravenous
Number analyzed (Participants) | 16 | 16
nanograms*hour/milliliter/milligram | 10256 [8964 to 11734] | 23150 [20234 to 26485]
Statistical Analysis 1: Comparison: Part B: LY2189265 Subcutaneous vs Part B: LY2189265 Intravenous; Test type: Superiority or Other; Mixed Linear effects model analyses; Ratio of Geometric LS Mean = 0.443, 90% CI 2-sided [0.395 to 0.497]

2. Primary Outcome: Maximum Concentration (Cmax) of LY2189265: Subcutaneous (SC) to Intravenous (IV)
Description: The results presented are Geometric Least Squares (LS) Mean. LS Mean values were controlled for participants, sequence, treatment, period and random error.
Time Frame: Predose up to 336 hours postdose
Population: Participants in Part B who had pharmacokinetic (PK) data.
Measure: Geometric Mean (90% Confidence Interval); unit: nanograms/milliliter (ng/mL)
Groups:
- Part B: LY2189265 Subcutaneous: Single 1.5-milligram (mg) subcutaneous (SC) dose of LY2189265 in Period 1 or 2
Arm/Group | Part B: LY2189265 Subcutaneous | Part B: LY2189265 Intravenous
Number analyzed (Participants) | 16 | 16
nanograms/milliliter (ng/mL) | 80.7 [71.8 to 90.8] | 38.3 [34.1 to 43.1]
Statistical Analysis 1: Comparison: Part B: LY2189265 Subcutaneous vs Part B: LY2189265 Intravenous; Test type: Superiority or Other; Mixed Linear effects model analyses; Ratio of Geometric LS Mean = 2.10, 90% CI 2-sided [1.84 to 2.41]

3. Secondary Outcome: Area Under the Concentration Time Curve (AUC) of LY2189265: Intramuscular (IM) to Subcutaneous (SC)
Description: as for outcome 1
Time Frame: Predose up to 336 hours postdose
Population: Participants in Part C who had pharmacokinetic (PK) data.
Measure: Geometric Mean (90% Confidence Interval); unit: nanograms*hour/milliliter (ng*h/mL)
Groups:
- Part C: LY2189265 Intramuscular: Single 0.75-milligram (mg) intramuscular (IM) of LY2189265 in Period 1or 2
- Part C: LY2189265 Subcutaneous: Single 0.75-mg subcutaneous (SC) dose of LY2189265 in Period 1 or 2
Arm/Group | Part C: LY2189265 Intramuscular | Part C: LY2189265 Subcutaneous
Number analyzed (Participants) | 7 | 8
nanograms*hour/milliliter (ng*h/mL) | 9828 [7525 to 12837] | 10215 [7832 to 13323]
Statistical Analysis 1: Comparison: Part C: LY2189265 Intramuscular vs Part C: LY2189265 Subcutaneous; Test type: Superiority or Other; Mixed Linear effects model analyses; Ratio of Geometric LS Means = 0.962, 90% CI 2-sided [0.858 to 1.08]

4. Secondary Outcome: )Maximum Concentration (Cmax) of LY2189265: Intramuscular (IM) to Subcutaneous (SC)
Description: as for outcome 2
Time Frame: Predose up to 336 hours postdose
Population: Participants in Part C who had pharmacokinetic (PK) data.
Measure: Geometric Mean (90% Confidence Interval); unit: nanograms/milliliter (ng/mL)
Groups:
- Part C: LY2189265 Intramuscular: Single 0.75-milligram (mg) intramuscular (IM) of LY2189265 in Period 1 or 2
Arm/Group | Part C: LY2189265 Intramuscular | Part C: LY2189265 Subcutaneous
Number analyzed (Participants) | 7 | 8
nanograms/milliliter (ng/mL) | 56.9 [48.4 to 67.0] | 54.2 [46.3 to 63.5]
Statistical Analysis 1: Comparison: Part C: LY2189265 Intramuscular vs Part C: LY2189265 Subcutaneous; Test type: Superiority or Other; Mixed Linear effects model analyses; Ratio of Geometric LS Means = 1.05, 90% CI 2-sided [0.924 to 1.19]

ADVERSE EVENTS:
Groups:
- Part A: 0.1 mg IV LY2189265: Single 0.1-milligram (mg) intravenous (IV) dose of LY2189265
- Part B: 0.1 mg IV LY2189265: Single 0.1-mg intravenous (IV) dose of LY2189265 in Period 1 or 2.
- Part B: 1.5 mg SC LY2189265: Single 1.5-mg subcutaneous (SC) dose of LY2189265 in Period 1 or 2.
- Part C: 0.75 mg IM LY2189265: Single 0.75-mg intramuscular (IM) of LY2189265 in Period 1 or 2.
- Part C: 0.75 mg SC LY2189265: Single 0.75-mg subcutaneous (SC) dose of LY2189265 in Period 1 or 2.
Arm/Group | Part A: 0.1 mg IV LY2189265 | Part B: 0.1 mg IV LY2189265 | Part B: 1.5 mg SC LY2189265 | Part C: 0.75 mg IM LY2189265 | Part C: 0.75 mg SC LY2189265
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/16 | 0/16 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/6 | 7/16 | 9/16 | 3/8 | 2/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: 0.1 mg IV LY2189265 (N=6) | Part B: 0.1 mg IV LY2189265 (N=16) | Part B: 1.5 mg SC LY2189265 (N=16) | Part C: 0.75 mg IM LY2189265 (N=8) | Part C: 0.75 mg SC LY2189265 (N=8)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 2 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Application site erythema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Extravasation (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oedema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site haematoma (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Procedural site reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 6 (7) | 1 (1) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days